CLINICAL TRIAL: NCT05547659
Title: Comparison Between Multimodal and Unimodal Analgesia in Cholecystectomy
Brief Title: Multimodal and Unimodal Analgesia in Cholecystectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, engy wahsh, head of clinical pharmacy unit, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA00015574
Record Dates: First submitted 2022-08-25; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Compare Unimodal and Multimodal Analgesics
MeSH Terms: interventions — Pregabalin; Acetaminophen; Tablets; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multimodal (Active Comparator): pregabalin/ acetaminophen/ celecoxib
  Interventions: Drug: Pregabalin 150mg; Drug: Acetaminophen 1 G Oral Tablet; Drug: Celecoxib 400Mg Oral Capsule
- unimodal (Active Comparator): Pregabalin
  Interventions: Drug: Pregabalin 150mg
- control (No Intervention)

INTERVENTIONS:
Drug: Pregabalin 150mg — Pregabalin 150mg preoperative in unimodal group Pregabalin 150mg preoperative in multi-modal group
  Arms: multimodal; unimodal
Drug: Acetaminophen 1 G Oral Tablet — Acetaminophen 1 G Oral Tablet preoperative in multi-modal group
  Arms: multimodal
Drug: Celecoxib 400Mg Oral Capsule — Celecoxib 400Mg Oral Capsule preoperative in multi-modal group
  Arms: multimodal

SUMMARY:
Many surgical procedures are accompanied by postoperative pain with severity moderate, severe or extreme and insufficient postoperative pain control may cause risk of post-surgical complications and risk of chronic post-surgical pain The targets of preoperative pain management are to relieve patient suffering, reduce length of hospital stay and achieve early mobilization after surgery, decreasing opioid consumption and its side effects that are constipation, nausea, vomiting, dizziness, respiratory depression which is the most feared complication being life-threatening and some less common side effects as sedation

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* Patients older than 18 years old

Exclusion Criteria:

* Renal or hepatic or cardiac impairment patients
* Patients with chronic pain history
* Allergic patients after taking aspirin or other NSAIDs
* patients with active gastrointestinal bleeding, ulcer and inflammatory bowel diseases or cerebrovascular bleeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative visual analogue scale (VAS) | 24 hour postoperative
  The visual analog scale (VAS) is a simple and often used method for evaluating variations in pain intensity.
Amount of post operative Needed opioid analgesia | 24 hour postoperative
  ampules of opioid analgesia needed after operation

SECONDARY OUTCOMES:
Type and amount of prescribed post operative non opioid analgesia | 24 hour postoperative
  Type and amount of prescribed post operative non opioid analgesia

OTHER OUTCOMES:
Reported opioid side effects | 24 hour postoperative
  Side effects reported after opioid administration eg. nausea, vomiting, respiratory depression etc..

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni suef University hospital, Banī Suwayf
  - Beni-Suef Hospital, Banī Suwayf

IPD SHARING:
Plan to Share IPD: Undecided